CLINICAL TRIAL: NCT02452892
Title: A Phase 2 Multicenter, Double-Blind, Placebo-Controlled, Dose Optimization Study of Low Field Magnetic Stimulation (LFMS) in Subjects With Treatment-Resistant Depression (TRD)
Brief Title: Low Field Magnetic Stimulation (LFMS) in Subjects With Treatment-Resistant Depression (TRD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tal Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAL-02-007
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-09

CONDITIONS: Depression; Depressive Disorder; Depressive Disorder, Treatment-resistant; Depressive Disorder, Major
Keywords: Depression; Major depression; Low-field magnetic stimulation; LFMS
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LFMS Sham (Sham Comparator): For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered. Low field magnetic stimulation (no magnetic field for sham) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  Interventions: Device: LFMS
- LFMS 20 minutes (Active Comparator): LFMS 20 minutes + Sham 40 min.Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  Interventions: Device: LFMS
- LFMS 60 minutes (Active Comparator): LFMS 60 minutes.Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  Interventions: Device: LFMS
- LFMS 120 min (Other): Week 2 subjects may be re-randomized to receive LFMS 120 minutes. Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  Interventions: Device: LFMS

INTERVENTIONS:
Device: LFMS — Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS. For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered.
  Other Names: Low Field Magnetic Stimulation

SUMMARY:
The purpose of this study is to compare the relative effectiveness of 20 and 60 minutes of Low-Field Magnetic Stimulation in relieving symptoms in patients with major depression who are treatment resistant.

DETAILED DESCRIPTION:
The primary objective of this study:

* To compare the relative efficacy, as measured by a change in the 6-item Hamilton Rating Scale for Depression (HAM-D6), of 20 and 60 minutes of LFMS compared to sham (placebo) in subjects with treatment resistant depression (TRD).

Secondary objectives:

* To determine if subjects with TRD may respond to 120 minutes of LFMS.
* To determine the persistence of response to LFMS therapy during the observation period.
* To evaluate the safety and tolerability of LFMS.

ELIGIBILITY:
Inclusion Criteria: (Key)

* Meets the Diagnostic and Statistical Manual of Mental Disorder, 5th Edition (DSM-5) criteria for Major Depressive Disorder (MDD), as determined by psychiatric evaluation.
* Has TRD of the current MDE, as assessed at the site by the Massachusetts General Hospital/Antidepressant Treatment Response Questionnaire (MGH/ATRQ).
* On an adequate dose of one antidepressant therapy (ADT) for at least eight weeks prior to the screening visit (Visit 1). The ADT dose must be stable for at least four weeks prior to the screening visit (Visit 1). Subjects must be willing to remain on the same stable dose of ADT upon signing the informed consent form until the end of the treatment observation period (end of Week 2) and, where possible, to the end of study participation

Exclusion Criteria: (Key)

* Have failed four or more lifetime adequate ADT treatment regimens (including the ongoing ADT for the current MDE).
* Have been treated with adjunctive antipsychotic medication with an antidepressant for at least two weeks during the current depressive episode.
* Are deemed to be at significant risk for suicidal behavior
* Are unable to lie on their back for the duration of study treatment
* Have a lifetime history of:

  1. Delirium, dementia, amnestic, or other cognitive disorder;
  2. Schizophrenia or any psychotic disorder, based on the Structured Clinical Interview for DSM-5 Axis I Disorders Patient Edition (SCID-I/P);
  3. Bipolar I or II disorder, based on the SCID-I/P.
* Have a current DSM-5 diagnosis at the screening visit (Visit 1) of:

  1. An eating disorder active within the 12 months prior to the screening visit (Visit 1);
  2. Comorbid anxiety disorders that predominate over MDD, as assessed by the investigator;
  3. Alcohol or substance use disorder active within the 12 months prior to the screening visit (Visit 1);
  4. Clinically significant DSM-5 Axis II disorder.
* Have ever received electroconvulsive therapy, vagal nerve stimulation, deep brain stimulation or repetitive transcranial magnetic stimulation.
* Have a non-removable programmable device or appliance such as cardiac pacemakers or cochlear implants.
* Have any non-removable ferromagnetic implants, or conductive or other magnetic sensitive materials present in the head or neck .
* Have a lifetime history of seizures or clinically significant electroencephalography abnormalities. A history of childhood febrile seizures is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Pande, MD, Study Chair — Tal Medical
Locations (12):
- United States (12):
  - CNS Trials, Garden Grove, California
  - Synergy Escondido, Lemon Grove, California
  - Pacific Trials Partners, Oakland, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - CNS Healthcare, Jacksonville, Florida
  - Segal Institute, Lauderhill, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Radiant Research, Atlanta, Georgia
  - Neurobehavioral-Clinical Research, Canton, Ohio
  - Midwest Clinical, Dayton, Ohio
  - Future Search Trials, Dallas, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12clinical study sites in the US recruited 122 subjects that were randomized into the study. The date of first subject enrollment was 03 September 2015 and the date of last subject enrolled was 22 July 2016.
Pre-assignment Details: Subject screening period was up to 14 days before receiving first study treatment. Subjects were contacted by an independent Massachusetts General Hospital-Clinical Trials Network and Institute (MGH-CTNI) rater to perform the Antidepressant Treatment Response Questionnaire (ATRQ) and SAFER assessments to confirm eligibility.
Groups:
- LFMS Sham: For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered.Week 1 subjects were randomly assigned using 1:1:1 allocation to LFMS Sham, LFMS 20 min., or LFMS 60 min. For Week 2 subjects were reassigned to LFMS Sham, LFMS 20min, LFMS 60min, or LFMS 120min. on the basis of their response to treatment received in Week 1 and their original treatment allocation.
- LFMS 20 Minutes: LFMS 20 minutes + Sham 40 min.Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  Week 1 subjects were randomly assigned using 1:1:1 allocation to LFMS Sham, LFMS 20 min., or LFMS 60 min. For Week 2, subjects were reassigned to LFMS Sham, LFMS 20min, LFMS 60min, or LFMS 120min. on the basis of their response to treatment received in Week 1 and their original treatment allocation.
- LFMS 60 Minutes: LFMS 60 minutes.Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  Week 1: Subjects were randomly assigned using 1:1:1 allocation to LFMS Sham, LFMS 20 min., or LFMS 60 min. For Week 2 subjects were reassigned to LFMS Sham, LFMS 20min, LFMS 60min, or LFMS 120min. on the basis of their response to treatment received in Week 1 and their original treatment allocation.
- LFMS 120 Min: Week 2: Subjects may be re-randomized to receive LFMS 120 minutes. Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  Week 1 subjects were randomly assigned using 1:1:1 allocation to LFMS Sham, LFMS 20 min., or LFMS 60 min. For Week 2 subjects were reassigned to LFMS Sham, LFMS 20min, LFMS 60min, or LFMS 120min. on the basis of their response to treatment received in Week 1 and their original treatment allocation.
Period: Week 1 Initial Randommization
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes | LFMS 120 Min
Started (Week 1 subjects were randomized 1:1:1 allocation to LFMS Sham, LFMS 20min,or LFMS 60min) | 41 | 40 | 41 | 0
Completed | 40 | 40 | 40 | 0
Not Completed | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Period: Week 2 Stratification & Re-Randomization
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes | LFMS 120 Min
Started (Subjects stratified by response & re-randomized to LFMS Sham, LFMS 20min, LFMS 60min, or LFMS 120min) | 65 (Week 1 Participants that started LFMS sham (27), LFMS 20min (19), and LFMS 60min (19)) | 7 (Week 1 Participants that Started LFMS Sham (0), LFMS 20min (7), and LFMS 60min(0).) | 7 (Week 1 Participants that Started LFMS Sham (0),LFMS 20min (0), LFMS 60min (7)) | 41 (Week 1 Participants that Started LFMS Sham (13), LFMS 20min (14), and LFMS 60 min (14).)
Non-reponders | 38 | 0 | 0 | 41
Responders | 27 | 7 | 7 | 0
Completed | 63 | 7 | 7 | 39
Not Completed | 2 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Period: Follow-up
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes | LFMS 120 Min
Started | 63 | 7 | 7 | 39
Completed | 62 | 7 | 7 | 38
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Subject left town on Day 42 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LFMS Sham: For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered. Low field magnetic stimulation (no magnetic field for sham) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  LFMS: Low field magnetic stimulation (1 kHz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS. For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered.
- LFMS 20 Minutes: LFMS 20 minutes + Sham 40 min.Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  LFMS: Low field magnetic stimulation (1 kHz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS. For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered.
- LFMS 60 Minutes: LFMS 60 minutes.Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  LFMS: Low field magnetic stimulation (1 kHz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS. For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered.
- LFMS 120 Min: Week 2 subjects may be re-randomized to receive LFMS 120 minutes. Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  LFMS: Low field magnetic stimulation (1 kHz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS. For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered.
- Total: Total of all reporting groups
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes | LFMS 120 Min | Total
Number analyzed (Participants) | 41 | 40 | 41 | 0 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 35 | 37 | 0 | 109
  >=65 years | 4 | 5 | 4 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 26 | 0 | 72
  Male | 18 | 17 | 15 | 0 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — White, Black or African American, Asian
  Participants
    White | 31 | 28 | 27 | 0 | 86
    Black or African American | 9 | 9 | 11 | 0 | 29
    Asian | 1 | 3 | 2 | 0 | 6
    Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to ( Day 4) in the 6-item Hamilton Rating Scale for Depression (HAM-D6) Total Score.
Description: Hamilton Rating Scales for Depression were designed to measure the severity of depressive symptoms in subjects with primary depressive illness. HAM-D6 is a subset of the HAM-D17 that assesses 6 items associated with major depression. The scale uses HAM-D17 items 1, 2, 7, 8, 10 and 13. Item 13 is scored 0 to 2 and all others are scored 0 to 4. Total score ranges from 0 to 22; higher score indicates more depression. Change from baseline: mean score at Week 1 Day 4 minus mean score at baseline".
  Week 1 Day 4 : Change from baseline to the end of the efficacy period ( Day 4) in the 6-item Hamilton Rating Scale for Depression (HAM-D6) total score .Responders at Day 4 will be defined as those subjects who achieve a decrease in HAM-D6 total score of 50% or more compared to baseline (Day 1, Week 1). All other subjects will be deemed to be non-responders at Day 4. Each patient's total score is his/her own reference for determining a decrease of 50% or more.
Time Frame: Week 1 Day 4
Population: Subjects in the All Randomized set who completed at least one treatment session and had at least one post baseline primary efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes
Number analyzed (Participants) | 41 | 40 | 41
units on a scale | -4.0 [-5.18 to -2.91] | -4.2 [-5.34 to -3.04] | -4.9 [-6.03 to -3.73]
Statistical Analysis 1: Comparison: LFMS Sham vs LFMS 60 Minutes; Comparisons of 60 min LFMS vs. sham, LSMean diff with 95% Confidence Interval (CI) reported. Hypothesis 1: no difference between 60 min. LFMS and sham therapy in mean change from baseline (Day 1) to end of Tx Day 4 in HAM-D6 total score. If hypothesis is rejected at significance level of 0.05, then second hypothesis will be tested. Hypothesis 2:no difference between 20 min. LFMS & sham therapy in mean change from baseline (Day 1) to the end of Tx. Day 4 in HAM-D6 total score; Test type: Superiority — To control for multiple comparisons in the primary endpoint analysis, a hierarchical approach was taken. First LFMS 60min. was compared to LFMS sham. If p<0.05 for this comparison, then LFMS 20min. was formally compared to LFMS sham for statistical significance; p = 0.307, Mixed Models Analysis — P-value displayed for 60min. Mixed Model Repeated Measures (MMRM) model; Week 1 baseline HAM-D6 total score, treatment,visit treatment*visit age, & gender included in model. Visit was the repeated measure within subjects
Statistical Analysis 2: Comparison: LFMS Sham vs LFMS 20 Minutes; Comparisons of 20 min LFMS vs. sham, LSMean diff with 95% Confidence Interval (CI) reported. Hypothesis 1: no difference between 60 min. LFMS and sham therapy in mean change from baseline (Day 1) to end of Tx Day 4 in HAM-D6 total score. If hypothesis is rejected at significance level of 0.05, then second hypothesis will be tested. Hypothesis 2:no difference between 20 min. LFMS & sham therapy in mean change from baseline (Day 1) to the end of Tx. Day 4 in HAM-D6 total score; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.859, Mixed Models Analysis — P-value displayed for 20min. Mixed Model Repeated Measures (MMRM) model; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Day 4 in HAM-D6 Total Score at Day 11 for Week 1 Non-responders: Response to 120 Minutes LFMS
Description: Hamilton Rating Scales for Depression were designed to measure the severity of depressive symptoms in subjects with primary depressive illness. HAM-D6 is a subset of the HAM-D17 that assesses 6 items associated with major depression. The scale uses HAM-D17 items 1, 2, 7, 8, 10 and 13. Item 13 is scored 0 to 2 and all others are scored 0 to 4. Total score ranges from 0 to 22; higher score indicates more depression. Change from Day 11: mean score at Week 2 Day 11 minus mean score at Day 4".
  To determine if subjects with TRD who are non-responders to 0, 20 or 60 minutes of LFMS on Day 4 may respond to 120 minutes of LFMS at the end of Day 11.
  Responders will be defined as those subjects who achieve a decrease in HAM-D6 total score of 50% or more compared to baseline (Day 1, Week 1). All other subjects will be deemed to be non-responders. Each patient's total score is his/her own reference for determining a decrease of 50% or more.
Time Frame: Day 11 (Week 2)
Population: Only non-responders at end of Day 4 comprise this Wk 2 analysis . (Non-responders were defined as those who didn't reach a decrease in 6-item Hamilton Rating Scale for Depression (HAM-D6) total score of 50% compared to baseline Day 1, Week 1). 41 subjects entered Week 2: 1 subject withdrew consent on Day 8 and was not part of the Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LFMS Sham | LFMS 120 Min
Number analyzed (Participants) | 38 | 40
units on a scale | -2.6 [-3.60 to -1.68] | -2.6 [-3.56 to -1.67]
Statistical Analysis 1: Comparison: LFMS Sham vs LFMS 120 Min; Test type: Superiority; p = 0.966, Mixed Models Analysis — P-value is not adjusted for multiple comparisons. P-value was estimated from Mixed Model Repeated Measures (MMRM) model; Week 2 baseline HAM-D6 total score, treatment, visit, treatment*visit, age, & gender included in model. Visit was the repeated measure within subject

3. Secondary Outcome: Day 4 Responders: Persistence of Effect Based on Pre-specified HAM-D6 Total Score
Description: To determine the persistence of response to LFMS therapy during a four-week follow-up period in subjects who were responders at Day 4. Persistence of response was achieved if during Week 2 post baseline visits and follow-up visits subjects' 6-item Hamilton Rating Scale for Depression (HAM-D6) total scores were lower than or equal to 50% of the baseline ( Day1 Week1) scores. Non-responder imputation method was used where missing post-baseline dichotomous ("yes or no") were imputed as non-responder. Logistic regression model used to compare treatment groups for each visit, where the model considers the treatment, age and gender as covariates.
Time Frame: Day 42
Population: Subjects who were HAM-D6 Day 4 responders, defined as those subjects who achieved a 50% or greater decrease in their HAM-D6 total score compared to Baseline ( Day1, Wk 1).
Measure: Number; unit: percentage of LFMS responders
Arm/Group | LFMS 20 Minutes | LFMS 60 Minutes | LFMS Sham
Number analyzed (Participants) | 13 | 14 | 14
percentage of LFMS responders | 53.8 | 57.1 | 78.6
Statistical Analysis 1: Comparison: LFMS 60 Minutes vs LFMS Sham; Test type: Superiority — The persistence rate calculated based on Week 1 treatment group: 20 minutes LFMS, 60 minutes LFMS and sham therapy; p = 0.294, Regression, Logistic — For 60 min LFMS, P-value not adjusted for multiple comparisons. P-value estimated using LR model including Wk2 baseline HAM-D6 total score, treatment, age & gender as covariates; Non-responder imputation (NRI) for missing data, where missing post-baseline results were considered non-response
Statistical Analysis 2: Comparison: LFMS 20 Minutes vs LFMS Sham; Test type: Superiority — The persistence rate calculated based on Week 1 treatment group: 20 minutes LFMS, 60 minutes LFMS and sham therapy; p = 0.232, Regression, Logistic — For 20min. LFMS, P-value not adjusted for multiple comparisons. P-value estimated using Logistic Regression model including Wk2 baseline HAM-D6 total score, treatment, age & gender as covariates; Non-responder imputation (NRI) for missing data, where missing post-baseline results were considered non-response

4. Post Hoc Outcome: Montgomery-Asberg Depression Rating Scale (MADRS): Change From Week 1 Baseline (Day 1) to End of Week 1 (Day 4)
Description: The MADRS is a 10-item checklist designed to measure the overall severity of depressive symptoms in subjects with Major Depressive Disorder (MDD). Individual items are rated on a scale of 0 to 6 in which a score of 6 represents the most severe symptoms for each item assessed. The total score ranges from 0 to 60.
  Remission of depression based on the MADRS is defined as a subject with a MADRS total score of ≤11 at endpoint. A responder on the MADRS is defined as a 50% or greater reduction from baseline in total MADRS score
Time Frame: Day 4 Week 1
Population: Full Analysis Set, Week1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes
Number analyzed (Participants) | 41 | 40 | 41
units on a scale | -7.58 [-9.8 to -5.4] | -8.09 [-10.3 to -5.8] | -10.32 [-12.6 to -8.0]
Statistical Analysis 1: Comparison: LFMS Sham vs LFMS 60 Minutes; Estimates for LS Means, confidence intervals, difference in LS means and p-value are from an ANCOVA model with treatment, age, sex as factors and baseline negative MADRS score as a covariate; Test type: Superiority; p = 0.0932, ANCOVA — P-value is not adjusted for multiple comparisons; P-value was estimated using ANCOVA model with treatment, age, & gender as factors and baseline negative MADRS score as a covariate
Statistical Analysis 2: Comparison: LFMS Sham vs LFMS 20 Minutes; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7509, ANCOVA — The p-value is not adjusted for multiple comparisons; [statistical method as in outcome 4, analysis 1]

5. Post Hoc Outcome: Positive and Negative Affect Schedule (PANAS): Change From Baseline at Day 4 in Positive Score
Description: The PANAS comprises two mood scales, one that measures positive affect and the other that measures negative affect. Used as a psychometric scale, the PANAS can show relationships between positive and negative affect with personality stats and traits. Descriptors are used to define their meanings. Subjects completing the PANAS are required to respond to a 20-item test using 5-point scale that ranges from very slightly or not at all (1) to extremely (5).To calculate the positive affect score, added scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores can range from 10-50, which higher scores representing higher levels of positive affect, or the extent to which the individual feels enthusiastic, active and alert.
Time Frame: Day 4 Week 1
Population: Full Analysis Set (Week 1).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes
Number analyzed (Participants) | 41 | 40 | 41
units on a scale | 1.67 [-0.29 to 3.62] | 3.62 [1.63 to 5.62] | 3.24 [1.23 to 5.26]
Statistical Analysis 1: Comparison: LFMS Sham vs LFMS 60 Minutes; Test type: Superiority — Positive score is the sum of 10 items: 1,3,5,9,10,12,14,16,17,19; p = 0.2672, ANCOVA — P-value not adjusted for multiple comparisons; P-value estimated using ANCOVA model with treatment,age,& gender as factors & baseline positive PANAS score as a covariate
Statistical Analysis 2: Comparison: LFMS Sham vs LFMS 20 Minutes; Test type: Superiority — Positive score is the sum of 10 items: 1,3,5,9,10,12,14,16,17,19; p = 0.1660, ANCOVA — P-value not adjusted for multiple comparisons; [statistical method as in outcome 5, analysis 1]

6. Post Hoc Outcome: Positive and Negative Affect Schedule (PANAS) Change From Baseline in Negative Score at Day 4
Description: The PANAS comprises two mood scales, one that measures positive affect and the other that measures negative affect. Subjects completing the PANAS are required to respond to a 20-item test using 5-point scale that ranges from very slightly or not at all (1) to extremely (5).Negative affect scores can be obtained by adding up scores for items 2, 4, 6, 7, 8, 11, 13, 15, 18 and 20. The negative affect score can range from 10 to 50, with lower scores representing lower level of negative affect, or the extent to which the individual feels aversive mood states and general distress.
  This analysis outcome treated Item #2 as random missing data.
Time Frame: Day 4, Week 1
Population: Full analysis set, Week 1.Item #2 was incorrectly listed as "Disinterested" instead of "Distressed".resulting in incorrect data for this item for the first 16 subjects. The PANAS data for the first 16 randomized subjects and in total 72 data points was identified and removed from the database. See stats analysis for further details.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes
Number analyzed (Participants) | 41 | 40 | 41
units on a scale | -2.27 [-4.20 to -0.34] | -3.57 [-5.55 to -1.59] | -5.32 [-7.31 to -3.33]
Statistical Analysis 1: Comparison: LFMS Sham vs LFMS 60 Minutes; Due to item #2 error, analyses were done in the following manner to check robustness: * All missing values including these 72 data points in item #2 were considered as random missing data (values posted in outcome measures). * The 72 data points were removed & the negative score for affected subjects & visits were not calculated. * The 72 data points were imputed using worst value imputation algorithm (using score =5 as extremely) while other random missing values imputed by average; Test type: Superiority — Negative score is sum of 10 items: 2,4,6,7,8,11,13,15,18,20; p = 0.0307, ANCOVA — P-value not adjusted for multiple comparisons. All missing values including the 72 data points in Item#2 were considered as random missing data; P-value estimated using ANCOVA model with treatment, age, & gender as factors & baseline negative PANAS score as a covariate
Statistical Analysis 2: Comparison: LFMS Sham vs LFMS 20 Minutes; Due to item #2 error, analyses were done in the following manner to check robustness: All missing values including these 72 data points in item #2 were considered as random missing data (values posted in outcome measures). The 72 data points were removed & the negative score for affected subjects & visits were not calculated. The 72 data points were imputed using worst value imputation algorithm (using score =5 as extremely) while other random missing values imputed by average; Test type: Superiority — Negative score is sum of 10 items: 2,4,6,7,8,11,13,15,18,20; p = 0.3537, ANCOVA — P-value not adjusted for multiple comparisons. All missing values including the 72 data points in Item#2 were considered as random missing data; [statistical method as in outcome 6, analysis 1]

7. Post Hoc Outcome: Positive and Negative Affect Schedule (PANAS) Change From Baseline in Negative Score at Day 4
Description: The PANAS comprises two mood scales, one that measures positive affect and the other that measures negative affect. Subjects completing the PANAS are required to respond to a 20-item test using 5-point scale that ranges from very slightly or not at all (1) to extremely (5).Negative affect scores can be obtained by adding up scores for items 2, 4, 6, 7, 8, 11, 13, 15, 18 and 20. The negative affect score can range from 10 to 50, with lower scores representing lower level of negative affect, or the extent to which the individual feels aversive mood states and general distress.
  This analysis outcome treated Incorrect Item #2 where Item #2 data was removed.
Time Frame: Day 4
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes
Number analyzed (Participants) | 41 | 40 | 41
units on a scale | -2.95 [-5.03 to -0.87] | -3.78 [-5.94 to -1.59] | -5.58 [-7.74 to -3.41]
Statistical Analysis 1: Comparison: LFMS Sham vs LFMS 60 Minutes; [analysis description as in outcome 6, analysis 2]; Test type: Superiority — Negative score is sum of 10 items: 2,4,6,7,8,11,13,15,18,20; p = 0.0848, ANCOVA — P-value not adjusted for multiple comparisons. All missing values including the 72 data points in Item#2 were treated where incorrect Item #2 data was removed; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: LFMS Sham vs LFMS 20 Minutes; [analysis description as in outcome 6, analysis 2]; Test type: Superiority — Negative score is sum of 10 items: 2,4,6,7,8,11,13,15,18,20; p = 0.5930, ANCOVA — [p-value comment as in outcome 7, analysis 1]; [statistical method as in outcome 6, analysis 1]

8. Post Hoc Outcome: Positive and Negative Affect Schedule (PANAS) Change From Baseline in Negative Score at End of Week 1, Day 4
Description: The PANAS comprises two mood scales, one that measures positive affect and the other that measures negative affect. Subjects completing the PANAS are required to respond to a 20-item test using 5-point scale that ranges from very slightly or not at all (1) to extremely (5).Negative affect scores can be obtained by adding up scores for items 2, 4, 6, 7, 8, 11, 13, 15, 18 and 20. The negative affect score can range from 10 to 50, with lower scores representing lower level of negative affect, or the extent to which the individual feels aversive mood states and general distress.
  This analysis outcome approach took Incorrect Item #2 and imputed using worst possible value.
Time Frame: Day 4, Week 1
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes
Number analyzed (Participants) | 41 | 40 | 41
units on a scale | -2.29 [-4.24 to -0.34] | -3.50 [-5.49 to -1.51] | -5.36 [-7.36 to -3.36]
Statistical Analysis 1: Comparison: LFMS Sham vs LFMS 60 Minutes; [analysis description as in outcome 6, analysis 2]; Test type: Superiority — Negative score is sum of 10 items: 2,4,6,7,8,11,13,15,18,20; p = 0.0307, ANCOVA — P-value not adjusted for multiple comparisons. All missing values including the 72 data points in Item#2 were treated where incorrect Item #2 data was imputed using worst possible value; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: LFMS Sham vs LFMS 20 Minutes; [analysis description as in outcome 6, analysis 2]; Test type: Superiority — Negative score is sum of 10 items: 2,4,6,7,8,11,13,15,18,20; p = 0.3907, ANCOVA — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: Day 1- Day 42. Treatment-emergent events for Week 1 was defined as any Adverse Event (AE) that began on or after Day 1 treatment until the end of Day 7. Treatment-emergent AEs for Week 2 was defined as any AE that began on or after the Day 8 treatment until the end of Day 15 (not including the follow-up phase).
Description: "# affected" for each tx group is the incidence count for each event occurring from Day 1-42. Day 8 Re-randomization per response to Wk 1 tx & original tx assignment creates a higher exposure to LFMS Sham in Week 2. The "# at risk" for each tx group is total number of unique subjects who received at least one dose of tx being summarized during either Wk 1 or Wk 2.
Groups:
- LFMS 120 Min - Week 2: Week 2 subjects may be re-randomized to receive LFMS 120 minutes. Low field magnetic stimulation (1 kilohertz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS.
  LFMS: Low field magnetic stimulation (1 kHz oscillating magnetic field) will be administered using a portable tabletop device capable of generating time-varying electromagnetic fields of LFMS. For sham therapy, the device will be on; however, no magnetic field stimulation will be delivered.
Arm/Group | LFMS Sham | LFMS 20 Minutes | LFMS 60 Minutes | LFMS 120 Min - Week 2
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/40 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/40 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 20/79 | 14/40 | 13/41 | 10/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LFMS Sham (N=79) | LFMS 20 Minutes (N=40) | LFMS 60 Minutes (N=41) | LFMS 120 Min - Week 2 (N=41)
Headche (Nervous system disorders) | 7 (10) | 6 (7) | 4 (4) | 4 (6)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head Discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (2)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gasrtoenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gasrtoenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infecrion (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hair disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was not powered for secondary measures. Statistical significance for group-wise comparisons wasn't expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No